CLINICAL TRIAL: NCT03594344
Title: Additional Hyperbaric Oxygen After Lower Extremity Amputation - A Randomized Controlled Trial
Brief Title: Additional Hyperbaric Oxygen After Lower Extremity Amputation
Acronym: AHOLEA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Diakonhjemmet Hospital (Other)
Responsible Party: Principal Investigator, Elisabeth Ellingsen Husebye, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017/1587
Record Dates: First submitted 2018-06-15; First posted 2018-07-20 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-09

CONDITIONS: Diabetes Mellitus; Claudication, Intermittent; Critical Limb Ischemia; Osteomyelitis; Amputation; Lower Extremity Ulcer; Diabetic Angiopathy; Diabetic Neuropathies; Diabetic Foot
Keywords: Diabetic foot; Diabetes; Lower extremity amputation; Hyperbaric oxygen therapy; HBOT
MeSH Terms: conditions — Diabetes Mellitus; Intermittent Claudication; Chronic Limb-Threatening Ischemia; Osteomyelitis; Leg Ulcer; Diabetic Angiopathies; Diabetic Neuropathies; Diabetic Foot | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyperbaric oxygen therapy (Experimental): 30 sessions of Hyperbaric oxygen therapy, 90min treatment at 2,4 ATA(atmosphere absolute) with 100% oxygen.First session must be given within 7 days after initial amputation. Treatment is given as outpatient treatment after discharge from hospital.
  Interventions: Procedure: Hyperbaric oxygen therapy
- Control group (No Intervention): Control group will be given standard of care with follow up at the outpatient clinic after discharge from hospital.

INTERVENTIONS:
Procedure: Hyperbaric oxygen therapy — Breathing 100% oxygen for 30+30+30 min at 2,4 ATA. in a multiplace hyperbaric chamber. Total of 30 sessions
  Arms: Hyperbaric oxygen therapy

SUMMARY:
This study evaluates the effect of additional hyperbaric oxygen therapy after lower extremity amputation. The patients will be randomized after amputation to either a treatment group receiving hyperbaric oxygen therapy, or control group.

DETAILED DESCRIPTION:
Hyperbaric oxygen therapy has been used to treat hard to heal wounds for decades. Amputation, especially distal lower extremity amputations have the same problem with healing and patients often need to be re-amputated more proximally. In these patients oxygen levels are often the decisive factor. Providing additional oxygen under hyperbaric conditions will increase tissue oxygen concentration sufficient for the amputation stump to heal. This will give the patients a more distal amputation with better condition for ambulation.

ELIGIBILITY:
Inclusion Criteria:

* Lower extremity amputation because of chronic wound, osteomyelitis, ischemia, necrosis.
* Fit to receive hyperbaric oxygen therapy determined by an anesthesiologist/Hyperbaric Medicine Physician.
* Able to cooperate and follow up appointments
* Included within 7 days after final surgery

Exclusion Criteria:

* Not fulfilling inclusion criteria
* Pregnancy
* Dementia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-07-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Intact skin with no abnormal openings at the site of primary amputation | 12 weeks
  Healed and intact skin at the site of primary amputation without need for more proximal amputation.Healed amputation is defined as epithelialization of the wound examined by a orthopedic surgeon. Level of primary amputation is decided by the surgeon. Planned 2-session amputation, for example Guillotine amputation with a final amputation later is considered being primary amputation. Healed primary amputation will be measured at 12 weeks.

SECONDARY OUTCOMES:
Intact skin with no abnormal openings at the site of amputation at 6 months | 6 months
  Healed and intact skin at the site of amputation at follow up 6 months. Healed amputation is defined as epithelialization of the wound examined by a orthopedic surgeon.
Intact skin with no abnormal openings at the site of amputation at 9 months | 9 months
  Healed and intact skin at the site of amputation at follow up 9 months. Will be assessed if the wound has not healed at 6 months. Healed amputation is defined as epithelialization of the wound examined by a orthopedic surgeon.
Intact skin with no abnormal openings at the site of amputation at 1 year | 12 months
  Healed and intact skin at the site of amputation at follow up at 1 year. Healed amputation is defined as epithelialization of the wound examined by a orthopedic surgeon.
Time to closed and intact skin at the site of amputation | 1 year
  Time to closed and intact skin at the site of amputation is the defined as how many weeks until complete healing of amputation. Healed amputation is defined as epithelialization of the wound examined by a orthopedic surgeon and no abnormal openings.
Reamputations | 1 year
  The total number of reamputations done within the follow-up period of 1 year.
Number of wound revision | 1 year
  The total numbers of surgical wound revision done in operating theater.
Days in hospital during follow up | 1 year
  Total number of days in hospital during 1 year follow up
Visual analog pain scale (VAS) | baseline
  Visual analog pain scale (VAS) is a measurement of pain intensity between 0 and 10. 0 = no pain, 10 = worst imaginable pain.
Visual analog pain scale (VAS) | 12 weeks
  Visual analog pain scale (VAS) is a measurement of pain intensity between 0 and 10. 0 = no pain, 10 = worst imaginable pain.
Visual analog pain scale (VAS) | 6 months
  Visual analog pain scale (VAS) is a measurement of pain intensity between 0 and 10. 0 = no pain, 10 = worst imaginable pain.
Visual analog pain scale (VAS) | 1 year
  Visual analog pain scale (VAS) is a measurement of pain intensity between 0 and 10. 0 = no pain, 10 = worst imaginable pain.
RAND 36-Item Short Form Health Survey | baseline
  RAND 36-Item Short Form Health Survey (SF-36) measures 8 health domains with the total of 36 questions. The domains are physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. There is also 1 question that measures change in self-perceived health.The question answers is translated to a number between 0 meaning worst selv-perceived health and 100 meaning the best possible quality of health.Each domain will be presented with a number between 0 and 100.
RAND 36-Item Short Form Health Survey | 12 weeks
  RAND 36-Item Short Form Health Survey (SF-36) measures 8 health domains with the total of 36 questions. The domains are physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. There is also 1 question that measures change in self-perceived health.The question answers is translated to a number between 0 meaning worst selv-perceived health and 100 meaning the best possible quality of health.Each domain will be presented with a number between 0 and 100.
RAND 36-Item Short Form Health Survey | 6 months
  RAND 36-Item Short Form Health Survey (SF-36) measures 8 health domains with the total of 36 questions. The domains are physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. There is also 1 question that measures change in self-perceived health.The question answers is translated to a number between 0 meaning worst selv-perceived health and 100 meaning the best possible quality of health.Each domain will be presented with a number between 0 and 100.
RAND 36-Item Short Form Health Survey | 1 year
  RAND 36-Item Short Form Health Survey (SF-36) measures 8 health domains with the total of 36 questions. The domains are physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. There is also 1 question that measures change in self-perceived health.The question answers is translated to a number between 0 meaning worst selv-perceived health and 100 meaning the best possible quality of health.Each domain will be presented with a number between 0 and 100.
Quality of Life in Neurological Disorders - Lower extremity function - Mobility Short form | baseline
  Quality of Life in Neurological Disorders (Neuro-QoL) - Lower extremity function - Mobility Short form measures lower extremity function with 8 items scoring from 1 unable to do, to 5 which is doing it without any difficulty. Scores will be presented as total points from 5-40.
Quality of Life in Neurological Disorders - Lower extremity function - Mobility Short form | 12 weeks
  Quality of Life in Neurological Disorders (Neuro-QoL) - Lower extremity function - Mobility Short form measures lower extremity function with 8 items scoring from 1 unable to do, to 5 which is doing it without any difficulty. Scores will be presented as total points from 5-40.
Quality of Life in Neurological Disorders - Lower extremity function - Mobility Short form | 6 months
  Quality of Life in Neurological Disorders (Neuro-QoL) - Lower extremity function - Mobility Short form measures lower extremity function with 8 items scoring from 1 unable to do, to 5 which is doing it without any difficulty. Scores will be presented as total points from 5-40.
Quality of Life in Neurological Disorders - Lower extremity function - Mobility Short form | 1 year
  Quality of Life in Neurological Disorders (Neuro-QoL) - Lower extremity function - Mobility Short form measures lower extremity function with 8 items scoring from 1 unable to do, to 5 which is doing it without any difficulty. Scores will be presented as total points from 5-40.
The Foot and Ankle Ability Measure (FAAM) | baseline
  The Foot and Ankle Ability Measure (FAAM) is a self-report outcome instrument developed to assess physical function for individuals with foot and ankle related impairments. FAAM contains 21 items that measure different functions. Each answer get a score from 0 to 4. The score total will be reported were 0 is the lowest and 84 is the highest possible score.
The Foot and Ankle Ability Measure (FAAM) | 12 weeks
  The Foot and Ankle Ability Measure (FAAM) is a self-report outcome instrument developed to assess physical function for individuals with foot and ankle related impairments. FAAM contains 21 items that measure different functions. Each answer get a score from 0 to 4. The score total will be reported were 0 is the lowest and 84 is the highest possible score.
The Foot and Ankle Ability Measure (FAAM) | 6 months
  The Foot and Ankle Ability Measure (FAAM) is a self-report outcome instrument developed to assess physical function for individuals with foot and ankle related impairments. FAAM contains 21 items that measure different functions. Each answer get a score from 0 to 4. The score total will be reported were 0 is the lowest and 84 is the highest possible score.
The Foot and Ankle Ability Measure (FAAM) | 1 year
  The Foot and Ankle Ability Measure (FAAM) is a self-report outcome instrument developed to assess physical function for individuals with foot and ankle related impairments. FAAM contains 21 items that measure different functions. Each answer get a score from 0 to 4. The score total will be reported were 0 is the lowest and 84 is the highest possible score.

CONTACTS AND LOCATIONS:
Overall Officials: Jonas V Rydinge, MD, Principal Investigator — Ullevål University Hospital, orthopedic department
Locations (2):
- Norway (2):
  - Diakonhjemmet Hospital, Oslo
  - Orthopedic Center, Ullevål University Hopspital, Oslo

IPD SHARING:
Plan to Share IPD: Undecided